CLINICAL TRIAL: NCT02121171
Title: Comparative Evaluation of Combined Trabeculotomy-trabeculectomy Versus Combined Trabeculotomy-trabeculectomy With Subconjunctival Implantation of Collagen Matrix Implant for Primary Congenital Glaucoma.
Brief Title: Combined Trab+Trab Versus Combined Trab+Trab With Subconjunctival Implantation of Ologen for Primary Congenital Glaucoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Centre of Ophthalmology named after academician Zarifa Aliyeva (Other Government)
Collaborators: Aeon Astron Europe B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Trab+Trab+Ologen
Record Dates: First submitted 2014-04-19; First posted 2014-04-23 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Congenital Glaucoma
MeSH Terms: conditions — Hydrophthalmos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ologen Collagen Matrix Intervention (Experimental): Combined trabeculotomy-trabeculectomy with subconjuncitval Ologen matrix implant implantation is a new procedure that has less post operative complications with good results, it is to be applied in children.
  Interventions: Device: Ologen Collagen Matrix
- Combined trabeculotomy-trabeculectomy (Active Comparator): Combined trabeculotomy and trabeculectomy is a standard surgery for congenital glaucoma, however, it has its known complications.
  Interventions: Procedure: Combined trabeculotomy-trabeculectomy

INTERVENTIONS:
Device: Ologen Collagen Matrix — Use of ologen Collagen Matrix in trabeculectomy (ologen) Place ologen CM on the top of the loosely-sutured scleral flap under conjunctiva before suturing. It is recommended to suture the scleral flap with 1 or 2 stiches loosely and to coordinate with the tamponading effect of ologen CM to create a fluctuating scleral flap that prevents bleb wound adhesion and modulates aqueous humor outflow for ideal IOP control without leakage.
  Arms: Ologen Collagen Matrix Intervention
Procedure: Combined trabeculotomy-trabeculectomy — Combined trabeculotomy and trabeculectomy is a standard surgery for congenital glaucoma, however, it has its known complications.
  Arms: Combined trabeculotomy-trabeculectomy

SUMMARY:
The objective of this prospective randomised study is to compare the efficacy and safety of ologen CM (Collagen matrix) as adjunct to combined trabeculotomy-trabecuectomy in congenital glaucoma cases, the efficacy being the primary objective and the safety being the secondary. The investigators hypothesize that combined trabeculotomy-trabecuectomy with Ologen collagen matrix implant implantation in congenital glaucoma is a safer procedure and may yield better results than combined trabeculotomy-trabeculectomy approach.

DETAILED DESCRIPTION:
"Ologen ® CM" is a biodegradable collagen matrix. To prevent episcleral fibrosis and subconjunctival scarring thay may result in the surgical failure in filtration surgery, its sporous matrix modulates the migrations and proliferations of fibroblasts to create a vascular and long-lasting bleb without the adverse effects.

Results of ologen CM studies have been published at conferences and published in peer-reviewed journals; ologen CM is approved in Europe as an aid for tissue repair, and by the FDA in the US as an adjunct in wound management(K080868). In general, over 7,000 ologen CM have been implanted worldwide during the past two years with good results and excellent safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Any case diagnosed as congenital glaucoma with enlarged corneal diameter more than 11 mm and intra-ocular pressure above 21 mmHg, including corneal edema or Haab's stria with or without optic disc cupping.

Any case diagnosed as primary or secondary congenital glaucoma to ocular or systemic abnormalities.

Within the age of (0 - 12).

Exclusion Criteria:

* Cases of congenital glaucoma with previous intervention. Age above 12 Yrs. Cases with secondary glaucoma caused by surgical intervention, ocular co-morbidity, medications or trauma

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2010-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure(IOP) reduction | At postoperative up to 24 months
  "Complete success" is consider for IOP less than 21mmHg(inclusive) with no glaucoma medications and with more than 20% reduction(inclusive) from baseline IOP.
  Definition of success rate is calculated in percentage by the number of complete success patients over the total sample size.
  "Qualified success" that meets the postoperative IOP requirements with postoperative glaucoma medicaitons and "Failure" of meeting the IOP requirements are the other efficacy parameters.
  In the specified time frame, patients will also visit for record at day 7, 30, 90, 180 days, 12, 18, and 24 months.

SECONDARY OUTCOMES:
Postoperative complications and appearances. | At postoperative up to 24 months.
  Inspections of hyphema, severe anterior chamber reaction, hypotony, supracholoidal hemorrhage, flat anterior chamber, endophthalmitis, choroidal detachment, wound or bleb leak.
  Visual acuity (if possible), bleb appearance, and anterior chamber inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Nigar Makhmudova, Principal Investigator — Ophthalmologist at National Centre of Ophthalmology
Locations (1):
- National Centre of Ophthalmology, Baku, Azerbaijan